CLINICAL TRIAL: NCT05540561
Title: Biological Alterations of Laughing Gas Outcomes in Neurology
Brief Title: Biological Diagnosis and Monitoring of Chronic Nitrous Oxide Abuse
Acronym: BALON
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2021_0461; 2022-A00327-36 (Other: 2022-A00327-36)
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-09

CONDITIONS: Nitrous Oxide Abuse
Keywords: Nitrous Oxide; Neurology; Thrombosis; Biomarkers; Metabolis
MeSH Terms: conditions — Thrombosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, serum, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects consuming nitrous oxide with clinical outcomes: Subjects who consume nitrous oxide and who have been hospitalized in this context and who present clinical signs determined during a neurological evaluation according to the PND (Peripheral Neuropathy Disability) score or who have had a thrombotic accident related to the consumption of nitrous oxide.
  Interventions: Other: blood collection
- Subjects consuming nitrous oxide without clinical outcomes: Subjects who consume nitrous oxide who do not present clinical signs related to this consumption and recruited during a routine medical consultation.
  Interventions: Other: blood collection

INTERVENTIONS:
Other: blood collection — Biological analyses in the framework of care with conservation of blood samples

SUMMARY:
There is a toxicity linked to the chronic use of nitrous oxide, leading to neurological disorders such as combined sclerosis of the spinal cord. One thus frequently observes patients presenting disorders of walking or paresthesias, of more or less resolving evolution being able to go until the need for using a wheelchair and more recently cases of thrombosis were reported Serum or urine N2O assays are rarely performed routinely, because they do not allow to ensure a real exposure due to the very short half-life of this gas in the body. Thus, other biological monitoring markers are mentioned in the literature, such as vitamin B12 or homocysteine. Unfortunately, there are still no recommendations for biological monitoring of nitrous oxide consumption. Moreover, underlying mechanisms leading to clinical outcomes remains misunderstood.

ELIGIBILITY:
Inclusion Criteria:

* A current or former recreational nitrous oxide user defined
* With associated clinical signs (group 1)
* Without associated clinical signs (group 2)
* With or without clinico-biological sequelae associated with use
* Consenting to the conduct of the study
* Socially insured

Exclusion Criteria:

* Pregnant or breastfeeding women
* Never used nitrous oxide or stopped using it more than 6 months ago
* Lack of social security coverage
* Not willing to participate in the entire study

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients using or having recently used nitrous oxide, and hospitalized during the study will be offered to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 356 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Blood markers related to nitrous oxide consumption | through study completion an average of 1 year
  Biomarkers of cobalamin metabolism, methionine cycle and oxidative stress

SECONDARY OUTCOMES:
Blood markers related to nitrous oxide clinical outcomes. | Baseline, at 4 weeks, at 3 months and at 6 months
  Biomarkers of cobalamin metabolism, methionine cycle and oxidative stress and biological markers of neurological damage.
Estimated and self-reported nitrous oxide consumption | Baseline, at 4 weeks,and/or at 3 months and at 6 months
The severity of the clinical signs related to nitrous oxide consumption. | Baseline, at 4 weeks,and/or at 3 months and at 6 months
  The severity of the signs noted during the interrogation and consultation of the patients by filling out a pre-established form listing the neurological signs (gait disorders evaluated by the PND score, presence of paresthesia and associated clinical signs (thrombotic and psychiatric events)

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - BETHUNE, Béthune
  - Boulogne Sur Mer, Boulogne-sur-Mer
  - CALAIS, Calais
  - Lens, Lens
  - Chu Lille, Lille
  - Nantes, Nantes
  - Roubaix, Roubaix
  - Rouen, Rouen